CLINICAL TRIAL: NCT03375632
Title: Clinical Pharmacological Study of FYU-981 Administered to Hyperuricemic Outpatients With or Without Gout
Brief Title: Study of FYU-981 in Hyperuricemic Outpatients With or Without Gout (Effect on Two Hyperuricemic Types)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mochida Pharmaceutical Company, Ltd. (Industry)
Collaborators: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FYU-981-013
Record Dates: First submitted 2017-12-10; First posted 2017-12-18 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Hyperuricemia With or Without Gout
MeSH Terms: interventions — dotinurad

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uric acid-overproduction Type (Experimental)
  Interventions: Drug: FYU-981
- Uric acid-underexcretion Type (Experimental)
  Interventions: Drug: FYU-981

INTERVENTIONS:
Drug: FYU-981 — Oral daily dosing for 14 weeks

SUMMARY:
To investigate the pharmacodynamics and safety of FYU-981 administered orally once a day for 14 weeks, to uric acid-overproduction type or uric acid-underexcretion type of male hyperuricemic outpatients with or without gout.

ELIGIBILITY:
Inclusion Criteria:

* Serum urate level:

  * >= 7.0mg/dL in patients with gouty nodule or with history of gout, or >=8.0mg/dL in patients with hypertension, diabetes or metabolic syndrome, or >= 9.0mg/dL
* Disease type in the classification of hyperuricemia: Uric acid-overproduction type or Uric acid-underexcretion type
* Outpatients

Exclusion Criteria:

* Gouty arthritis within 14 days before randomized allocation

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics (Amount of uric acid excreted in urine) | 2-week
Pharmacodynamics (Amount of uric acid excreted in urine) | 6-week
Pharmacodynamics (Amount of uric acid excreted in urine) | 10-week
Pharmacodynamics (Amount of uric acid excreted in urine) | 14-week

CONTACTS AND LOCATIONS:
Overall Officials: Kazuki Furuno, Study Director — Clinical Research Department
Locations (1):
- Mochida Investigational sites, Tokyo, Japan